CLINICAL TRIAL: NCT01894152
Title: Evaluate the Continued Safety and Effectiveness of the XIENCE PRIME EECSS in a Cohort of Real-world Patients Receiving the XIENCE PRIME EECSS During Commercial Use.
Brief Title: XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS) China Single-Arm Study
Acronym: XP China SAS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-396
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Angioplasty; Cardiovascular Disease; Coronary Artery Disease; Coronary Heart Disease; Coronary Restenosis; Myocardial Infarction; Stent Thrombosis; Vascular Disease
Keywords: XIENCE PRIME EECSS; XIENCE V EECSS; XIENCE PRIME; SPIRIT PRIME; XIENCE PRIME SV (Small Vessel); XIENCE PRIME LL (Long Lesion); Coronary Artery Disease; Coronary Heart Disease; Cardiovascular Disease; Myocardial Infarction; Stent Thrombosis
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease; Coronary Restenosis; Myocardial Infarction; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS): Subjects receiving XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
  Interventions: Device: XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)

INTERVENTIONS:
Device: XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS) — Subjects receiving XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)

SUMMARY:
Abbott Vascular (AV) obtained marketing approval for the XIENCE PRIME Everolimus Eluting Coronary Stent System (XIENCE PRIME EECSS) in China from the China Food and Drug Administration (CFDA) on August 10th, 2011.

This prospective, observational, open-label, multi-center, single-arm, post-approval study is designed to evaluate the continued safety and effectiveness of the XIENCE PRIME EECSS in a cohort of real-world patients receiving the XIENCE PRIME EECSS during commercial use in real-world settings in China.

This study has no primary outcome measure. All observations are of equal weight.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age at the time of signing the informed consent.
* The patient or his/her legally-authorized representative signs the European Commission (EC)-approved Informed Consent Form (ICF).
* Only XIENCE PRIME stent(s) is (are) implanted during the index procedure.

Exclusion Criteria:

* No other exclusion criteria are specified for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of real-world patients receiving the XIENCE PRIME EECSS during commercial use in realworld settings in China.
Sampling Method: Non-Probability Sample
Enrollment: 2002 (Actual)
Dates: Start 2013-07; Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MB, MSc, MD, Principal Investigator — Fudan University; Fang Chen, MD, Principal Investigator — Anzhen Hospital
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2140 patients were registered from 35 centres in China. First patients was enrolled on July 12, 2013 & enrollment was completed on Sep11, 2014 through the Interactive Voice Response System (IVRS) excluding those without consent and those without stent implants & duplicate entries. Thus the analysis population includes 2002 participants .
Pre-assignment Details: Of the 2140 registered subjects,138 subjects withdrew from the study due to incomplete consent forms, no implanted study stents and repeated entry in voice interactive selection system. Among the final analysis population (n=2002), a total of 151 subjects failed to complete the follow-up period.
Period: Overall Study
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Started | 2002
Completed | 1851
Not Completed | 151
Not completed — No DMR and no Stent thrombosis | 151

BASELINE CHARACTERISTICS:
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 2002
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1286
  >=65 years | 716
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.42 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 501
  Male | 1501
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2002
Region of Enrollment [Count of Participants; unit: Participants]
  China | 2002

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cardiac Death and All Myocardial Infarction (MI) (Q-wave and Non-Q Wave) Composite Endpoint
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded.
  (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality, cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.)
  Myocardial Infarction (MI):
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of Creatine kinase (CK) levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: Full Analysis Set (FAS). Full Analysis Set includes all patients who had implanted XIENCE PRIME EECSS stent in the start-up procedures. The analysis population includes patients with DMR composite event (deaths, myocardial infarctions, revascularization cases) or stent thrombosis or complete follow-up at given point in time.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 7

2. Other Pre Specified Outcome: Number of Participants With Cardiac Death and All Myocardial Infarction (MI) (Q-wave and Non-Q Wave) Composite Endpoint
Description: as for outcome 1
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 114

3. Other Pre Specified Outcome: Number of All Deaths, Myocardial Infarction, Any Repetitive Revascularization Composite Endpoints
Description: All deaths include Cardiac death, Cardiovascular death and Non-cardiovascular death.
  Myocardial Infarction (MI):
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of Creatine kinase (CK) levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 8

4. Other Pre Specified Outcome: Number of All Deaths, Myocardial Infarction, Any Repetitive Revascularization Composite Endpoints
Description: as for outcome 3
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 330

5. Other Pre Specified Outcome: Number of Participants With Cardiogenic Death, Target Vessel Blood Flow Myocardial Infarction, Target Lesion Revascularization Composite Endpoint
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded.
  (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality, cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.)
  Myocardial Infarction (MI): Patient diagnosed with myocardial infarction, but its relation with target vessel not clear, therefore considered target vessel myocardial infarction.
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of Creatine kinase (CK) levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 5

6. Other Pre Specified Outcome: Number of Participants With Cardiogenic Death, Target Vessel Blood Flow Myocardial Infarction, Target Lesion Revascularization Composite Endpoint
Description: as for outcome 5
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 120

7. Other Pre Specified Outcome: Number of Participants With Composite Rate of All Deaths and Myocardial Infarctions (MI)
Description: as for outcome 3
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 8

8. Other Pre Specified Outcome: Number of Participants With Composite Rate of All Deaths and Myocardial Infarctions (MI)
Description: as for outcome 3
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 156

9. Other Pre Specified Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Target Lesion Failure is composite of Cardiac death/ Target Vessel Myocardial Infarction (TV-MI)/ Ischemic-Driven Target Lesion Revascularization (ID-TLR).
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 5

10. Other Pre Specified Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 9
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 100

11. Other Pre Specified Outcome: Number of Participants With Target Vessel Failure (ID-TVF) (Cardiac Death, All Myocardial Infarctions and Ischemia-driven Target Vessel Revascularization)
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or ischemia-driven Target Vessel Revascularization (ID-TVR).
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 7

12. Other Pre Specified Outcome: Number of Participants With Target Vessel Failure (ID-TVF) (Cardiac Death, All Myocardial Infarctions and Ischemia-driven Target Vessel Revascularization)
Description: as for outcome 11
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 180

13. Other Pre Specified Outcome: Number of All Death (Cardiac, Vascular, and Non-cardiovascular)
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.) This study as no primary or secondary endpoints, all endpoints are of equal weight.
  - Non-cardiac death is defined as a death not due to cardiac causes (as defined above).
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 3

14. Other Pre Specified Outcome: Number of All Death (Cardiac, Vascular, and Non-cardiovascular)
Description: as for outcome 13
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 91

15. Other Pre Specified Outcome: Number of Participants With All Myocardial Infarction (MI) (Including Q-wave and Non-Q-wave)
Description: Myocardial Infarction (MI)
  * Q wave MI Development of new, pathological Q wave on the ECG
  * Non-Q wave MI Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 6

16. Other Pre Specified Outcome: Number of Participants With All Myocardial Infarction (MI) (Including Q-wave and Non-Q-wave)
Description: as for outcome 15
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 75

17. Other Pre Specified Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: Target Vessel Revascularization is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
  This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 0

18. Other Pre Specified Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 17
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 26

19. Other Pre Specified Outcome: Number of Participants With All Revascularization (Target Lesion, Target Vessel, and Non-target Vessel) (PCI and Coronary Artery Bypass Graft [CABG])
Description: This study has no primary or secondary endpoints, all endpoints are of equal weight.
  All Revascularization includes Coronary artery bypass grafting and Percutaneous coronary intervention
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 1

20. Other Pre Specified Outcome: Number of Participants With All Revascularization (Target Lesion, Target Vessel, and Non-target Vessel) (PCI and Coronary Artery Bypass Graft [CABG])
Description: as for outcome 19
Time Frame: 0 through 1885 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 223

21. Other Pre Specified Outcome: Number of Participants With Acute Stent Thrombosis
Description: This study has no primary or secondary endpoints, all endpoints are of equal weight.
  Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Acute scaffold/stent thrombosis : 0 - 24 hours post stent implantation Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation Extremely late scaffold/stent thrombosis: >1 year post stent implantation"
Time Frame: 0 to 1 day
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 0

22. Other Pre Specified Outcome: Number of Participants With Sub-acute Stent Thrombosis
Description: as for outcome 21
Time Frame: > 1 day to 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 2

23. Other Pre Specified Outcome: Number of Participants With Early Stent Thrombosis
Description: as for outcome 21
Time Frame: 0 - 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 2

24. Other Pre Specified Outcome: Number of Participants With Late Stent Thrombosis
Description: as for outcome 21
Time Frame: 31 to 365 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 1

25. Other Pre Specified Outcome: Number of Participants With Very Late Stent Thrombosis
Description: as for outcome 21
Time Frame: > 365 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 0

26. Other Pre Specified Outcome: Number of Participants With Overall Stent Thrombosis
Description: as for outcome 21
Time Frame: 0 to 1885 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 3

27. Other Pre Specified Outcome: Number of Participants With Target Vessel ARC MI
Description: This study has no primary or secondary endpoints, all endpoints are of equal weight.
  Myocardial Infarction (MI):
  Q wave MI: Development of new, pathological Q wave on the ECG. Non-Q wave MI: Elevation of Creatine kinase (CK) levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 2

28. Other Pre Specified Outcome: Number of Participants With Target Vessel ARC MI
Description: as for outcome 27
Time Frame: 0 to 1885 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 23

29. Other Pre Specified Outcome: Number of Participants With All TVR (TLR and TVR, Non-target Lesion)
Description: This study has no primary or secondary endpoints, all endpoints are of equal weight.
  All TVR (TLR and TVR, non-target lesion)
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 1

30. Other Pre Specified Outcome: Number of Participants With All TVR (TLR and TVR, Non-target Lesion)
Description: as for outcome 29
Time Frame: 0 to 1885 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 84

31. Other Pre Specified Outcome: Number of Participants With All TLR
Description: This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 1

32. Other Pre Specified Outcome: Number of Participants With All TLR
Description: This study has no primary or secondary endpoints, all endpoints are of equal weight.
Time Frame: 0 to 1885 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 58

33. Other Pre Specified Outcome: Number of Participants With ID-TLR
Description: This study has no primary or secondary endpoints, all endpoints are of equal weight.
  Revascularization includes TLR, TVR, non-target lesion, and non TVR.
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 1

34. Other Pre Specified Outcome: Number of Participants With ID-TLR
Description: as for outcome 33
Time Frame: 0 to 1885 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 37

35. Other Pre Specified Outcome: Number of Participants With ID-TVR, Non-target Lesion
Description: as for outcome 33
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 0

36. Other Pre Specified Outcome: Number of Participants With ID-TVR, Non-target Lesion
Description: as for outcome 33
Time Frame: 0 to 1885 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 22

37. Other Pre Specified Outcome: Number of Participants With ID-TVR (TLR and TVR, Non-target Lesion)
Description: as for outcome 33
Time Frame: ≤ 7 days after index procedure (Hospitalization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 1

38. Other Pre Specified Outcome: Number of Participants With ID-TVR (TLR and TVR, Non-target Lesion)
Description: as for outcome 33
Time Frame: 0 to 1885 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
Number analyzed (Participants) | 1851
Participants | 59

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS)
All-Cause Mortality (participants affected / at risk) | 91/2002
Serious Adverse Events (participants affected / at risk) | 1105/2002
Other Adverse Events (participants affected / at risk) | 103/2002
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS) (N=2002)
ANEMIA (Blood and lymphatic system disorders) | 1
BLOOD DISEASE (Blood and lymphatic system disorders) | 1
MASSIVE ABDOMINAL HEMORRHAGE (Blood and lymphatic system disorders) | 1
CHEST PAIN-CARDIAC (Cardiac disorders) | 16
CHEST PAIN AND CHEST TIGHTNESS (CHD) (Cardiac disorders) | 4
ACUTE CORONARY SYNDROME (Cardiac disorders) | 7
ACUTE HEART FAILURE (Cardiac disorders) | 3
ACUTE NON - ST SEGMENT ELEVATION MYOCARDIAL INFARCTION (Cardiac disorders) | 6
ACUTE ST-SEGMENT ELEVATION MYOCARDIAL INFARCTION (Cardiac disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 49
UNSTABLE ANGINA PECTORIS (Cardiac disorders) | 169
CHEST TIGHTNESS-CARDIAC (Cardiac disorders) | 9
ARRHYTHMIA (Cardiac disorders) | 10
ARRHYTHMIA PERMANENT PACEMAKER IMPLANTATION (Cardiac disorders) | 1
ARRHYTHMIA, ATRIAL FIBRILLATION (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 13
ATRIAL FLUTTER (Cardiac disorders) | 2
ATRIAL PREMATURE BEAT (Cardiac disorders) | 1
VENTRICULAR PREMATURE BEAT (Cardiac disorders) | 3
CORONARY HEART DISEASE (Cardiac disorders) | 236
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC DYSFUNCTION (Cardiac disorders) | 1
CARDIAC ENLARGEMENT (Cardiac disorders) | 1
CARDIAC INSUFFICIENCY (Cardiac disorders) | 1
CARDIAC RESPIRATORY ARREST (Cardiac disorders) | 1
CARDIAC TAMPONADE (Cardiac disorders) | 1
CHRONIC CORONARY INSUFFICIENCY (Cardiac disorders) | 1
HEART FAILURE (Cardiac disorders) | 24
CONGENITAL ATRIAL SEPTAL DEFECT (Cardiac disorders) | 1
CORONARY ATHEROSCLEROTIC CARDIOPATHY (Cardiac disorders) | 13
CORONARY HEART DISEASE DEATH (Cardiac disorders) | 2
EXTRASYSTOLE (Cardiac disorders) | 1
HEART PALPITATIONS (Cardiac disorders) | 1
HYDROPERICARDIUM (Cardiac disorders) | 2
ISCHEMIC CARDIOMYOPATHY (Cardiac disorders) | 3
LETHAL MYOCARDIAL INFARCTION (Cardiac disorders) | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 66
OLD MYOCARDIAL INFARCTION (Cardiac disorders) | 7
MYOCARDIAL BRIDGE (Cardiac disorders) | 1
NON-TARGET VESSEL REVASCULARIZATION (Cardiac disorders) | 5
PRECORDIAL DISTRESS (Cardiac disorders) | 2
SICK SINUS SYNDROME (Cardiac disorders) | 1
TACHYCARDIA-BRADYCARDIA SYNDROME (Cardiac disorders) | 1
TARGET LESION REVASCULARIZATION (Cardiac disorders) | 1
TRANSIENT ISCHEMIC ATTACK (Cardiac disorders) | 1
TVR or TLR (Cardiac disorders) | 21
VENTRICULAR FIBRILLATION (Cardiac disorders) | 2
CHRONIC HEART FAILURE (Cardiac disorders) | 1
BINOCULAR CATARACT (Eye disorders) | 1
LEFT EYE SENILE CATARACT (Eye disorders) | 1
RIGHT EYE CATARACT (Eye disorders) | 1
TRACTIONAL RETINAL DETACHMENT (Eye disorders) | 1
RIGHT EYE SENILE CATARACT (MATURE PERIOD) (Eye disorders) | 1
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 8
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 19
BLACK STOOL (Gastrointestinal disorders) | 1
CHRONIC GASTRITIS (Gastrointestinal disorders) | 2
CHRONIC NON-ATROPHIC GASTRITIS WITH BILE REFLUX (Gastrointestinal disorders) | 1
CHRONIC NON-ATROPHIC GASTRITIS WITH EROSION (Gastrointestinal disorders) | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1
GASTRIC ULCER WITH BLEEDING (Gastrointestinal disorders) | 3
LEFT INGUINAL HERNIA (Gastrointestinal disorders) | 1
CHEST PAIN (General disorders) | 58
CHEST PAIN AND CHEST TIGHTNESS (General disorders) | 8
CHEST TIGHTNESS (General disorders) | 63
BREASTBONE HIND TIGHTENING FEELING (General disorders) | 1
CHEST BLEEDING (General disorders) | 1
CHEST DISCOMFORT (General disorders) | 3
CHEST DISTRESS (General disorders) | 7
CHEST HEART PALPITATIONS (General disorders) | 1
DEATH (General disorders) | 42
DISCOMFORT IN THE ANTERIOR REGION OF THE HEART (General disorders) | 1
DIZZY (General disorders) | 4
EDEMA (General disorders) | 1
INTERMITTENT CHEST DISCOMFORT (General disorders) | 1
SYNCOPE (General disorders) | 5
MULTI-ORGAN FAILURE (General disorders) | 1
NECK DISCOMFORT (General disorders) | 1
PALPITATION (General disorders) | 9
THE AREA BEFORE THE HEART PALPITATIONS, SHORTNESS (General disorders) | 1
THE AREA BEFORE THE HEART TIGHTNESS (General disorders) | 1
THE LIMBS SWELLING (General disorders) | 1
TO TREAT OTHER VASCULAR LESIONS (General disorders) | 1
VERTIGO SYNDROME (General disorders) | 1
WEAK (General disorders) | 1
ACUTE PANCREATITIS (Hepatobiliary disorders) | 1
CONSTRICTIVE PERICARDITIS (Hepatobiliary disorders) | 1
HEMORRHAGE OF LIVER (Hepatobiliary disorders) | 1
LIVER FAILURE (Hepatobiliary disorders) | 2
NON-TARGET VESSEL PCI (Injury, poisoning and procedural complications) | 1
PCI POSTOPERATIVE UPPER GASTROINTESTINAL BLEEDING (Injury, poisoning and procedural complications) | 1
POSTOPERATIVE PCI (Injury, poisoning and procedural complications) | 1
REVASCULARIZATION (Injury, poisoning and procedural complications) | 7
REVASCULARIZATION OF LCX (Injury, poisoning and procedural complications) | 1
REVIEW AFTER PCI (Injury, poisoning and procedural complications) | 1
STENT THROMBOSIS (Injury, poisoning and procedural complications) | 3
STENT RESTENOSIS (Injury, poisoning and procedural complications) | 1
TOXIC MULTIPLE NEUROPATHY CAUSED BY DRUG (Injury, poisoning and procedural complications) | 1
CORONARY HEART DISEASE AND POST- PCI (Investigations) | 3
CORONARY HEART DISEASE REEXAMINATION (Investigations) | 2
CORONORY ANGIOGRAPHY(NOS) (Investigations) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 3
DIABETIC KETOACIDOSIS CAUSE THE DEATH (Metabolism and nutrition disorders) | 1
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2
HYPERTHYREOSIS (Metabolism and nutrition disorders) | 1
GOUT (Musculoskeletal and connective tissue disorders) | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
CANCER OF THE STOMACH (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CANCER METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
DESCENDING COLON TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ESOPHAGEAL MALIGNANT TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LIVER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LIVER CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATIC HYPERPLASIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PULMONARY HEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SACRAL TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
STOMACH CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BILATERAL OVARIAN CYSTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ACUTE BRAINSTEM INFARCTION (Nervous system disorders) | 1
ANGIONEUROEDEMA (Nervous system disorders) | 1
CEREBRAL INSUFFICIENCY (Nervous system disorders) | 1
CERVICAL HEADACHE (Nervous system disorders) | 1
DEATH(CEREBRAL INFARCTION AND CEREBRAL HERNIA) (Nervous system disorders) | 1
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 1
ISCHEMIC CEREBROVASCULAR DISEASE (Nervous system disorders) | 1
LACUNAR INFARCTION (Nervous system disorders) | 2
LEFT TEMPORAL LOBE BRAIN CONTUSION (Nervous system disorders) | 1
LUMBAR SPINAL STENOSIS (Nervous system disorders) | 1
STROKE (Nervous system disorders) | 1
SUBARACHNOID HEMORRHAGE (Nervous system disorders) | 1
BILATERAL URETERAL CALCULI (Renal and urinary disorders) | 2
RENAL FAILURE (Renal and urinary disorders) | 2
RIGHT HYDRONEPHROSIS WITH URETERAL STRICTURE (Renal and urinary disorders) | 1
ENDOMETRIAL LESIONS (Reproductive system and breast disorders) | 1
OOPHORITIC CYST (Reproductive system and breast disorders) | 1
VAGINAL BLEEDING (Reproductive system and breast disorders) | 1
BRONCHIAL ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 5
ANHELATION (Respiratory, thoracic and mediastinal disorders) | 2
CHEST TIGHTNESS AND SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 2
COPD (Respiratory, thoracic and mediastinal disorders) | 1
LEFT PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
LUNG INFECTION (Respiratory, thoracic and mediastinal disorders) | 2
MAXILLARY SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1
MIXED LUNG VENTILATION DYSFUNCTION (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 5
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY INFECTION (Respiratory, thoracic and mediastinal disorders) | 3
PULMONARY MULTILOBE PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
SEVERE PNEUMONIA AND RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
TYPE I RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
LACERATION OF SCALP SOFT TISSUE (Skin and subcutaneous tissue disorders) | 1
ABDOMINAL ANEURYSM (Vascular disorders) | 1
ABNORMAL VESSELS IN CORONARY ARTERIES (Vascular disorders) | 1
ARTERIOSCLEROSIS OBLITERANS OF LOWER EXTREMITY (Vascular disorders) | 1
ATHEROSCLEROSIS (Vascular disorders) | 1
CAROTID ARTERY OCCLUSION (Vascular disorders) | 1
CEREBRAL HEMORRHAGE (Vascular disorders) | 7
CEREBRAL INFARCTION (Vascular disorders) | 12
HYPERTENSION (Vascular disorders) | 7
INSUFFICIENT BLOOD SUPPLY TO THE CEREBRAL ARTERY (Vascular disorders) | 1
POSTERIOR CIRCULATION ISCHEMIA (Vascular disorders) | 5
PULMONARY EMBOLISM (Vascular disorders) | 1
SEQUELAE OF CEREBRAL INFARCTION (Vascular disorders) | 2
VASCULAR STENOSIS (Vascular disorders) | 1
VENTRICULAR ANEURYSM (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE PRIME Everolimus Eluting Coronary Stent System (EECSS) (N=2002)
HEMORRHOIDAL BLEEDING (Blood and lymphatic system disorders) | 2
ANGINA PECTORIS (Cardiac disorders) | 10
AURICULAR FIBRILLATION (Cardiac disorders) | 1
CHEST PAIN - CARDIAC (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 3
HEART FAILURE (Cardiac disorders) | 2
MI (Cardiac disorders) | 2
PREMATURE BEAT (Cardiac disorders) | 2
REPERFUSION ARRHYTHMIA (Cardiac disorders) | 2
RESTING ANGINA (Cardiac disorders) | 1
UNSTABLE ANGINA (Cardiac disorders) | 10
BLEEDING IN EYES (Eye disorders) | 3
DEFECATE HAEMORRHAGE (Gastrointestinal disorders) | 2
GASTRIC COLIC (Gastrointestinal disorders) | 1
GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 8
UPSET STOMACH (Gastrointestinal disorders) | 2
BLEEDING (General disorders) | 1
BLEEDING GUMS (General disorders) | 6
CHEST PAIN (General disorders) | 5
CHEST TIGHTEN AND CARDIOPALMUS (General disorders) | 1
CHEST TIGHTNESS (General disorders) | 4
DIZZY (General disorders) | 1
FEEL SUFFOCATED (General disorders) | 1
HEMORRHAGIC SPOT (General disorders) | 1
PALPITATION (General disorders) | 3
SHORT OF BREATH (General disorders) | 1
STOMACHACHE (General disorders) | 1
SYNCOPE (General disorders) | 1
TOOTHACHE (General disorders) | 1
(General disorders) | 1
OM1 SEGMENT OCCLUDED (Injury, poisoning and procedural complications) | 1
CNI IS HIGHER THAN NORMAL VALUE (Investigations) | 1
ELEVATED TROPOLIN T (Investigations) | 3
ELEVATED TROPONIN I (Investigations) | 6
LACUNAR INFARCTION (Nervous system disorders) | 1
VAGAL REFLEX (Nervous system disorders) | 1
VERTEBRAL STENOSIS (Nervous system disorders) | 1
NOSE BLEEDING (Respiratory, thoracic and mediastinal disorders) | 2
SUBCUTANEOUS HEMORRHAGE (Skin and subcutaneous tissue disorders) | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 1
SKIN ALLERGY (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-05-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT01894152/SAP_000.pdf
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT01894152/Prot_001.pdf